CLINICAL TRIAL: NCT07000617
Title: A Phase II Study of Dexamethasone, Azacitidine, Pegaspargase and Tislelizumab Plus Radiotherapy for Patients With Stage I/II Extranodal NK/T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University International Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1-2151
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: NK/T Cell Lymphoma
Keywords: NK/T cell lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DAPT regimen plus radiotherapy (Experimental): Patients receive 6 cycles of DAPT regimen plus concurrent radiotherapy. The DAPT regimen consists of dexamethasone, azacitidine, pegaspargase and tislelizumab.
  Interventions: Drug: DAPT regimen plus radiotherapy

INTERVENTIONS:
Drug: DAPT regimen plus radiotherapy — Patients receive 6 cycles of DAPT regimen plus concurrent radiotherapy. The DAPT regimen is administered as follows: dexamethasone 10mg intravenously on days1-3, azacitidine 100mg subcutaneously on days 1-5, pegaspargase 2500IU/m2 intramuscularly on day 1, and tislelizumab 200mg intravenously on day 6, repeated every 21 days. Concurrent radiotherapy given to the tumor sites is started after 2 cycles of DAPT regimen. The specific doses and methods of radiotherapy are in accordance with the clinical guidelines for NK/T-cell lymphoma.

SUMMARY:
The goal of this clinical trial is to learn if the regimen of dexamethasone, azacitidine, pegaspargase and tislelizumab (DAPT regimen) combined with radiotherapy works to treat stage I or II NK/T cell lymphoma in adults. It will also learn about the safety of the DAPT regimen. The main questions it aims to answer are:

What are the efficacy of the DAPT regimen plus radiotherapy in participants with extranodal NK/T-cell lymphoma? What medical problems do participants have when taking the DAPT regimen?

Participants will:

Receive the DAPT regimen every 21 days for 6 cycles and radiotherapy Visit the clinic according to clinical trial requirement for checkups and tests Receive blood tests and radiological imaging tests according to the clinical trial requirement

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of extranodal NK/T-cell lymphoma
2. Age ≥18 years
3. Ann Arbor stage I or II
4. Presence of at least 1 measurable lesion according to the 2014 Lugano revised criteria for response assessment
5. ECOG-PS 0~2
6. Peripheral blood absolute neutrophil count ≥1.5×10E9/L, platelet count ≥75×10E9/L and hemoglobin ≥90g/L
7. Expected survival of at least 3 months
8. Capable of understanding the content of this study, agreeing to participate in this study and signing the informed consent.

Exclusion Criteria:

1. Unconfirmed pathological diagnosis of NK/T-cell lymphoma
2. Pregnant or lactating women, or patients of childbearing age unwilling to take contraceptive measures during the study period.
3. Patients with clinically significant prolonged QTc interval (>470ms in males, >480ms in females), ventricular tachycardia, atrial fibrillation, second or third degree atrioventricular block, acute myocardial infarction, congestive heart failure, severe or symptomatic coronary artery disease requiring medical treatment.
4. Patients with large amount of pericardial effusions shown by echocardiogram.
5. Patients who received supportive care for anemia, neutropenia or thrombocytopenia within 7 days prior to start of study treatment.
6. Patients with severe active bleeding.
7. Patients with pulmonary embolism, intracranial hemorrhage or acute cerebral infarction.
8. Patients with active infectious disease.
9. Patients who are mentally disabled or unable to understand or sign the informed consent form.
10. Patients with other conditions judged as ineligible for this study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | From enrollment to the end of treatment at 8 weeks
  Complete response rate is assessed according to the 2014 Lugano criteria for response assessment of lymphoma.

SECONDARY OUTCOMES:
Objective response rate | From enrollment to the end of treatment at 8 weeks
  Objective response rate is assessed according to the 2014 Lugano criteria for response assessment of lymphoma, including complete response and partial response.
2-year progression-free survival rate | From enrollment to 2 years after the end of treatment
  Progression-free survival (PFS) is measured from the time of start of treatment to the time of first progression, relapse after response, death from any cause, or the date of last follow-up. 2-year PFS rate will be estimated using the Kaplan-Meier method.
2-year overall survival rate | From enrollment to 2 years after the end of treatment
  Overall survival (OS) is defined as the time from the start of treatment to the time of death from any cause or the date of last follow-up. The 2-year OS rate will be estimated using the Kaplan-Meier method.
Adverse events | From enrollment to the end of treatment at 1 month
  All adverse events will be recorded and graded according to CTCAE 5.0

OTHER OUTCOMES:
Exploratory biomarker analyses | From enrollment to 2 years after the end of treatment
  Patients' tumor tissue and blood samples will be collected and analyzed to explore predictive biomarkers for treatment response and prognosis.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - National Cancer Center / Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - Peking University Cancer Hospital, Beijing
  - Peking University International Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided